CLINICAL TRIAL: NCT00215410
Title: Study in Patients With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Director, Clinical Affairs, Dey
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DL-055
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2008-02

CONDITIONS: Asthma
Keywords: Asthma; Formoterol; Fumarate
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate

INTERVENTIONS:
Drug: Formoterol Fumarate

SUMMARY:
The purpose of this study is to determine the most safe and effective dose of the investigational drug in comparison with a control drug and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Children with a history of asthma
* Written guardian approval

Exclusion Criteria:

* Current or recent asthma exacerbation, requiring hospitalization
* History of smoking
* Debilitating or systemic and/or life-threatening diseases.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36
Dates: Primary Completion 2003-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Measure of lung function

SECONDARY OUTCOMES:
Change in lung function, as well as vital signs
Physical Exam results, AE reporting, etc

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Research Site, Little Rock, Arkansas
  - Research Site, Long Beach, California
  - Research Site, Mission Viejo, California
  - Research Site, Newport Beach, California
  - Research Site, Orange, California
  - Research Site, Vista, California
  - Research Site, Englewood, Colorado
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas